CLINICAL TRIAL: NCT00001832
Title: Treatment of Patients With Metastatic Melanoma Using Cloned Lymphocytes Following the Administration of a Non-Myeloablative But Lymphocyte Depleting Regimen
Brief Title: Lymphocyte Re-infusion During Immune Suppression to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, Dr. Steven Rosenberg, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990158; 99-C-0158; NCT00019942 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Immunotherapy; Adoptive Transfer; IL-2; Toxicity; Clinical Response; Breast Cancer
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Breast Neoplasms | interventions — montanide ISA 51; Interleukin-2; fludarabine; fludarabine phosphate; Cyclophosphamide; Filgrastim; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Abl Cells in culture (Experimental): Peripheral blood mononuclear cells (PBMC) and/or tumor infiltrating lymphocytes (TIL) obtained by apheresis or lesion excision to be cloned and expanded in the lab.The patients underwent an apheresis and/or an excision of their tumor.
  They didn't receive any drugs.
  Interventions: Procedure: Apheresis
- Abl Cells IV + Cyclophosphamide 30 mg/kg (Experimental): Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x30mg/kg + Cells intravenous (IV) Abl cells intravenous (IV) = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV + Cyclophosphamide 60 mg/kg (Experimental): Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV+Low Dose IV IL-2 (Initial) (Experimental): Phase 1 interleukin-2 (IL-2) Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV IL-2 (72,000 IU/kg q8h for a maximum of 15 doses) Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV+High Dose IV IL-2 (Initial) (Experimental): Phase 1 interleukin-2 (IL-2) Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV + MTD IL-2 (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF) (to shorten time to neutrophil recovery) Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IA + MTD (prior cells IV on 6) (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) Prior Cells IV + growth colony stimulating factor (G-CSF) Abl cells IA = Lymphocytes 10^9-10^11 IA over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IA + MTD IL-2 (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF) Abl cells IA = Lymphocytes 10^9-10^11 IA over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IA+MTD IL-2 (MART-1 reactive) (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF) + melanoma- associated antigen recognized by T cells (MART-1):26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells Abl cells IA = Lymphocytes 10^9-10^11 IA over 30 minutes on day 0, repeated in 14 to 21 days gp100 = gp100:209-217(210M) peptide - 1 mg in IFA SQ (in the subcutaneous tissue of each thigh) on the morning of the cell infusion, plus gp100:209-217(210M) peptide, 1 mg, in IFA injected into the subcutaneous tissue in two equal volumes, 1.0 mL for each injection, within 2cm of each other, in the thigh daily for five days starting on the morning of the cell infusion and then weekly for 3 more injections.
  Interventions: Drug: Montanide ISA-51; Drug: MART-1:26-35(27L); Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IV + MTD IL-2 no GCSF (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) without growth colony stimulating factor (G-CSF) (to determine if G-CSF has harmful effects when adoptively transferring lymphocytes following a nonmyeloablative chemotherapy regimen) Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV+MTD IL-2 no GCSF (Experimental): Abl Cells intravenous (IV) + maximum tolerated dose (MTD) interleukin-2 (IL-2) no growth colony stimulating factor (GCSF)(gp100 reactive).
  Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + gp100:209-217(210M) 1mg/day (2-8 days) in patients with gp100 reactive cells Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: gp100:209-217 (210M); Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV+MTD IL-2 (Experimental): Abl Cells intravenous (IV)+ maximum tolerated dose (MTD) interleukin-2 (IL-2) no growth colony stimulating factor (GCSF) (melanoma-associated antigen recognized by T cells (MART-1)reactive).
  Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Drug: MART-1:26-35(27L); Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Abl Cells IV + SQ IL-2 with GCSF (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + growth colony stimulating factor (G-CSF) (to shorten time to neutrophil recovery), reactivity not specified Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IV + SQ (Experimental): Abl Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) with growth colony stimulating factor (GCSF) (melanoma-associated antigen recognized by T cells (MART-1) reactive) Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Drug: MART-1:26-35(27L); Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)
- Abl Cells IV + SQ IL-2 with GCSF (no reactivity) (Experimental): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 ( IL-2) (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + growth colony stimulating factor (G-CSF) in patients with no reactivity Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days
  Interventions: Drug: IL-2; Biological: Abl cells; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCSF (Growth colony stimulating factor)

INTERVENTIONS:
Drug: gp100:209-217 (210M) — gp100 = gp100:209-217(210M) peptide - 1 mg in IFA SQ (in the subcutaneous tissue of each thigh) on the morning of the cell infusion, plus gp100:209-217(210M) peptide, 1 mg, in IFA injected into the subcutaneous tissue in two equal volumes, 1.0 mL for each injection, within 2cm of each other, in the thigh daily for five days starting on the morning of the cell infusion and then weekly for 3 more injections.
  MART-1 = MART-1:26-35(27L) peptide- 1 mg in IFA SQ (in the subcutaneous tissue of each thigh) on the morning of the cell infusion, plus MART-1:26-35(27L) peptide, 1 mg, in IFA injected into the subcutaneous tissue in two equal volumes, 1.0 mL for each injection, within 2cm of each other, in the thigh daily for five days starting on the morning of the cell infusion and then weekly for 3 more injections.
  Arms: Abl Cells IV+MTD IL-2 no GCSF
Drug: Montanide ISA-51 — MART-1 = MART-1:26-35(27L) peptide- 1 mg in IFA SQ (in the subcutaneous tissue of each thigh) on the morning of the cell infusion, plus MART-1:26-35(27L) peptide, 1 mg, in IFA injected into the subcutaneous tissue in two equal volumes, 1.0 mL for each injection, within 2cm of each other, in the thigh daily for five days starting on the morning of the cell infusion and then weekly for 3 more injections.
  Other Names: IFA
  Arms: Abl Cells IA+MTD IL-2 (MART-1 reactive)
Drug: IL-2 — 125,000 IU/kg dose intravenous for 5 days for 6 weeks with 2 days rest per week.
  720,000 IU/kg intravenous every 8 hours for a maximum of 12 doses.
  Other Names: Interleukin-2
  Arms: Abl Cells IA + MTD (prior cells IV on 6); Abl Cells IA + MTD IL-2; Abl Cells IV + MTD IL-2 no GCSF; Abl Cells IV + SQ; Abl Cells IV + SQ IL-2 with GCSF; Abl Cells IV + SQ IL-2 with GCSF (no reactivity); Abl Cells IV+High Dose IV IL-2 (Initial); Abl Cells IV+Low Dose IV IL-2 (Initial); Abl Cells IV+MTD IL-2; Abl Cells IV+MTD IL-2 no GCSF
Drug: MART-1:26-35(27L) — MART-1 = MART-1:26-35(27L) peptide- 1 mg in IFA SQ (in the subcutaneous tissue of each thigh) on the morning of the cell infusion, plus MART-1:26-35(27L) peptide, 1 mg, in IFA injected into the subcutaneous tissue in two equal volumes, 1.0 mL for each injection, within 2cm of each other, in the thigh daily for five days starting on the morning of the cell infusion and then weekly for 3 more injections.
  Other Names: melanoma-associated antigen recognized by T cells
  Arms: Abl Cells IA+MTD IL-2 (MART-1 reactive); Abl Cells IV + SQ; Abl Cells IV+MTD IL-2
Biological: Abl cells — Abl cells IV = Lymphocytes 10^9-10^11 IV over 30 minutes on day 0, repeated in 14 to 21 days Abl cells IA = Lymphocytes 10^9-10^11 IA over 30 minutes on day 0, repeated in 14 to 21 days
  Arms: Abl Cells IA + MTD (prior cells IV on 6); Abl Cells IA + MTD IL-2; Abl Cells IA+MTD IL-2 (MART-1 reactive); Abl Cells IV + Cyclophosphamide 30 mg/kg; Abl Cells IV + Cyclophosphamide 60 mg/kg; Abl Cells IV + MTD IL-2; Abl Cells IV + MTD IL-2 no GCSF; Abl Cells IV + SQ; Abl Cells IV + SQ IL-2 with GCSF; Abl Cells IV + SQ IL-2 with GCSF (no reactivity); Abl Cells IV+High Dose IV IL-2 (Initial); Abl Cells IV+Low Dose IV IL-2 (Initial); Abl Cells IV+MTD IL-2; Abl Cells IV+MTD IL-2 no GCSF
Drug: Fludarabine — 5x25 mg/m^2 intravenous
  Other Names: Fludara
  Arms: Abl Cells IA + MTD (prior cells IV on 6); Abl Cells IA + MTD IL-2; Abl Cells IA+MTD IL-2 (MART-1 reactive); Abl Cells IV + Cyclophosphamide 30 mg/kg; Abl Cells IV + Cyclophosphamide 60 mg/kg; Abl Cells IV + MTD IL-2; Abl Cells IV + MTD IL-2 no GCSF; Abl Cells IV + SQ; Abl Cells IV + SQ IL-2 with GCSF; Abl Cells IV + SQ IL-2 with GCSF (no reactivity); Abl Cells IV+High Dose IV IL-2 (Initial); Abl Cells IV+Low Dose IV IL-2 (Initial); Abl Cells IV+MTD IL-2; Abl Cells IV+MTD IL-2 no GCSF
Drug: Cyclophosphamide — 2x30 mg/kg, 2x60 mg/kg intravenous
  Other Names: Cytoxan
  Arms: Abl Cells IA + MTD (prior cells IV on 6); Abl Cells IA + MTD IL-2; Abl Cells IA+MTD IL-2 (MART-1 reactive); Abl Cells IV + Cyclophosphamide 30 mg/kg; Abl Cells IV + Cyclophosphamide 60 mg/kg; Abl Cells IV + MTD IL-2; Abl Cells IV + MTD IL-2 no GCSF; Abl Cells IV + SQ; Abl Cells IV + SQ IL-2 with GCSF; Abl Cells IV + SQ IL-2 with GCSF (no reactivity); Abl Cells IV+High Dose IV IL-2 (Initial); Abl Cells IV+Low Dose IV IL-2 (Initial); Abl Cells IV+MTD IL-2; Abl Cells IV+MTD IL-2 no GCSF
Biological: GCSF (Growth colony stimulating factor) — Beginning on day 1 or 2, GCSF will be administered subcutaneously at a dose of 5mcg/kg/day (not to exceed 300 mcg/day. Filgrastim administration will continue daily until neutrophil count > 1.0 x10^9/L x 3 days or > 5.0 x10^9/L.
  Other Names: Filgrastim
  Arms: Abl Cells IA + MTD (prior cells IV on 6); Abl Cells IA + MTD IL-2; Abl Cells IA+MTD IL-2 (MART-1 reactive); Abl Cells IV + MTD IL-2; Abl Cells IV + SQ; Abl Cells IV + SQ IL-2 with GCSF; Abl Cells IV + SQ IL-2 with GCSF (no reactivity)
Procedure: Apheresis
  Arms: Abl Cells in culture

SUMMARY:
This experiment will test the safety and effectiveness of a treatment for melanoma in which certain lymphocytes (a type of white blood cell) are taken from the patient, grown in the laboratory, and returned after the patient's immune system has been weakened with immune-suppressing drugs. Some patients will also receive interleukin-2 (IL-2), a drug that may enhance the activity of the re-infused lymphocytes.

Patients with metastatic melanoma (melanoma whose tumor has spread) who have been treated unsuccessfully with gp100 vaccination may participate in this study. They will undergo apheresis or a tumor biopsy, or both, to collect lymphocytes. In apheresis, whole blood is drawn through a needle in the arm. A machine separates the blood components and removes the white cells. The rest of the blood is returned to the donor through a needle in the other arm. A biopsy is a surgical procedure to remove a small piece of tumor tissue.

Several weeks before the lymphocytes are collected, patients will receive injections of growth colony stimulating factor (G-CSF) every day for five days. This drug stimulates white cell production, permitting as many cells as possible to be obtained during collection. The lymphocytes will then be grown in larger numbers in the laboratory.

Seven days before the cells are re-infused, the patient is admitted to the hospital and a catheter (small tube) is placed in a large vein in the chest or neck. Two drugs, cyclophosphamide and fludarabine, are given through the tube. These drugs suppress the immune system so that it will not interfere with the work of the reinfused lymphocytes. The lymphocytes are then injected through the catheter over a 30-minute period. After the infusion, patients who receive IL-2 will be given the drug in a high dose over a 15-minute period every eight hours for up to five days. Patients whose condition does not permit high-dose IL-2, such as those with a heart condition or lung problem, may receive a low-dose regimen, with the drug given as a shot under the skin of the thigh or abdomen for five days followed by a 2-day break, continuing for a total of six weeks. These patients receive a higher dose the first week and then half that dose the next five weeks.

Blood and tissue samples will be taken before and during the study to evaluate the size of the tumor and assess treatment. If, 3-5 weeks after therapy is completed, the patient's tumor has stabilized or shrunk, the entire treatment, except for chemotherapy, may be repeated two more times.

DETAILED DESCRIPTION:
Patients with metastatic melanoma who are human immunodeficiency virus (HIV) and Hepatitis B negative and who have previously progressed after receiving standard therapy will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine and then will be treated by the adoptive transfer of lymphocytes reactive with shared antigens on their tumors. This study will evaluate the toxicity, immunologic effects and potential therapeutic role of this treatment.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patients must have evaluable metastatic melanoma that is refractory to standard therapy.
* Age greater than or equal to 16 years.
* Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1 at entry to the trial and at the time of chemotherapy induction.
* Absolute neutrophil count greater than 1000/mm^3.
* Platelet count greater than 100,000/mm^3.
* Hemoglobin greater than 8.0 g/dl.
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than two times the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 1.6 mg/dl, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior therapy at the time the patient receives the preparative regimen.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* Life expectancy of greater than three months.
* No steroid therapy required.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen.
* Patients to receive high dose interleukin 2 (IL-2) must have no active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system.
* Patients who will receive high dose IL-2 as part of the phase I portion of this study or who will be randomized must be eligible to receive high dose IL-2.
* Any patient receiving IL-2 must sign a durable power of attorney.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1999-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Derived] Yao X, Ahmadzadeh M, Lu YC, Liewehr DJ, Dudley ME, Liu F, Schrump DS, Steinberg SM, Rosenberg SA, Robbins PF. Levels of peripheral CD4(+)FoxP3(+) regulatory T cells are negatively associated with clinical response to adoptive immunotherapy of human cancer. Blood. 2012 Jun 14;119(24):5688-96. doi: 10.1182/blood-2011-10-386482. Epub 2012 May 3. PMID 22555974
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_1999-C-0158.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Abl Cells in Culture: Peripheral blood mononuclear cells (PBMC) and/or tumor infiltrating lymphocytes (TIL) obtained by apheresis or lesion excision to be cloned and expanded in the lab. All patients were enrolled on Arm 0 and their cells were then sent to the lab. If the lab was able to manufacture the cell product then the patient was enrolled on one of the treatment arms.
- Abl Cells IV + Cyclophosphamide 30 mg/kg: Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x30mg/kg + Cells intravenous (IV)
- Abl Cells IV + Cyclophosphamide 60 mg/kg: Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV)
- Abl Cells IV+Low Dose IV IL-2 (Initial): Phase 1 interleukin-2 (IL-2) Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV IL-2 (72,000 IU/kg q8h for a maximum of 15 doses)
- Abl Cells IV+High Dose IV IL-2 (Initial): Phase 1 interleukin-2 (IL-2) Dose Escalation: Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses)
- Abl Cells IV + MTD IL-2: Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF) (to shorten time to neutrophil recovery)
- Abl Cells IA + MTD (Prior Cells IV on 6): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) Prior Cells IV + growth colony stimulating factor (G-CSF)
- Abl Cells IA + MTD IL-2: Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF)
- Abl Cells IA+MTD IL-2 (MART-1 Reactive): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intra-arterial (IA) + intravenous (IV) interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) + growth colony stimulating factor (G-CSF) + melanoma- associated antigen recognized by T cells (MART-1):26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Abl Cells IV + MTD IL-2 no GCSF: Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) without growth colony stimulating factor (G-CSF) (to determine if G-CSF has harmful effects when adoptively transferring lymphocytes following a nonmyeloablative chemotherapy regimen)
- Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive): Abl Cells intravenous (IV) + maximum tolerated dose (MTD) interleukin-2 (IL-2) no growth colony stimulating factor (GCSF)(gp100 reactive).Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + gp100:209-217(210M) 1mg/day (2-8 days) in patients with gp100 reactive cells
- Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive): Abl Cells intravenous (IV)+ maximum tolerated dose (MTD) interleukin-2 (IL-2) no growth colony stimulating factor (GCSF) (melanoma-associated antigen recognized by T cells (MART-1)reactive).Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV interleukin-2 (IL-2) (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Abl Cells IV + SQ IL-2 With GCSF: Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + growth colony stimulating factor (G-CSF) (to shorten time to neutrophil recovery), reactivity not specified
- Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive): Abl Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) with growth colony stimulating factor (GCSF) (melanoma-associated antigen recognized by T cells (MART-1) reactive) Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Abl Cells IV + SQ IL-2 With GCSF (no Reactivity): Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 ( IL-2) (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + growth colony stimulating factor (G-CSF) in patients with no reactivity
Period: Apheresis Period
Arm/Group | Abl Cells in Culture | Abl Cells IV + Cyclophosphamide 30 mg/kg | Abl Cells IV + Cyclophosphamide 60 mg/kg | Abl Cells IV+Low Dose IV IL-2 (Initial) | Abl Cells IV+High Dose IV IL-2 (Initial) | Abl Cells IV + MTD IL-2 | Abl Cells IA + MTD (Prior Cells IV on 6) | Abl Cells IA + MTD IL-2 | Abl Cells IA+MTD IL-2 (MART-1 Reactive) | Abl Cells IV + MTD IL-2 no GCSF | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) | Abl Cells IV + SQ IL-2 With GCSF | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity)
Started | 170 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 110 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — not able to manufacture treatment cells | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Abl Cells in Culture | Abl Cells IV + Cyclophosphamide 30 mg/kg | Abl Cells IV + Cyclophosphamide 60 mg/kg | Abl Cells IV+Low Dose IV IL-2 (Initial) | Abl Cells IV+High Dose IV IL-2 (Initial) | Abl Cells IV + MTD IL-2 | Abl Cells IA + MTD (Prior Cells IV on 6) | Abl Cells IA + MTD IL-2 | Abl Cells IA+MTD IL-2 (MART-1 Reactive) | Abl Cells IV + MTD IL-2 no GCSF | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) | Abl Cells IV + SQ IL-2 With GCSF | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity)
Started | 0 | 3 | 3 | 3 | 6 | 51 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2
Completed | 0 | 3 | 3 | 3 | 6 | 50 | 4 | 6 | 8 | 6 | 1 | 7 | 6 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death during treatment | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cells IV + Cyclophosphamide 30mg/kg: Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x30mg/kg + Cells IV
- Cells IV + Cyclophosphamide 60mg/kg: Phase 1 Cyclophosphamide Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV
- Cells IV + Low-Dose IV IL-2 (Initial): Phase 1 IL-2 Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (72,000 IU/kg q8h for a maximum of 15 doses)
- Cells IV + High-Dose IV IL-2 (Initial): Phase 1 IL-2 Dose Escalation: Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses)
- Cells IV + MTD IL-2: Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) + G-CSF (to shorten time to neutrophil recovery)
- Cells IA + MTD IL-2 (Prior Cells IV on 6): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IA + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) Prior Cells IV + G-CSF
- Cells IA + MTD IL-2: Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IA + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) + G-CSF
- Cells IA + MTD IL-2 (MART-1 Reactive): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IA + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) + G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Cells IV + MTD IL-2 no GCSF: Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF (to determine if G-CSF has harmful effects when adoptively transferring lymphocytes following a nonmyeloablative chemotherapy regimen)
- Cells IV + MTD IL-2 no GCSF (gp100 Reactive): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + gp100:209-217(210M) 1mg/day (2-8 days) in patients with gp100 reactive cells
- Cells IV + MTD IL-2 no GCSF (MART-1 Reactive): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + IV IL-2 (720,000 IU/kg q8h for a maximum of 12 doses) without G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Cells IV + SQ IL-2 w/GCSF: Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF (to shorten time to neutrophil recovery), reactivity not specified
- Cells IV + SQ IL-2 w/GCSF (MART-1 Reactive): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
- Cells IV + SQ IL-2 w/GCSF (no Reactivity): Phase 2 Fludarabine 5x25mg/m2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF in patients with no reactivity
- Total: Total of all reporting groups
Arm/Group | Cells IV + Cyclophosphamide 30mg/kg | Cells IV + Cyclophosphamide 60mg/kg | Cells IV + Low-Dose IV IL-2 (Initial) | Cells IV + High-Dose IV IL-2 (Initial) | Cells IV + MTD IL-2 | Cells IA + MTD IL-2 (Prior Cells IV on 6) | Cells IA + MTD IL-2 | Cells IA + MTD IL-2 (MART-1 Reactive) | Cells IV + MTD IL-2 no GCSF | Cells IV + MTD IL-2 no GCSF (gp100 Reactive) | Cells IV + MTD IL-2 no GCSF (MART-1 Reactive) | Cells IV + SQ IL-2 w/GCSF | Cells IV + SQ IL-2 w/GCSF (MART-1 Reactive) | Cells IV + SQ IL-2 w/GCSF (no Reactivity) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 51 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 3 | 3 | 3 | 5 | 51 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 1 | 108
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (9.3) | 52.3 (4.5) | 42.3 (13.3) | 37.8 (14.7) | 41.9 (12.7) | 38.0 (14.3) | 39.7 (11.1) | 41.8 (11.6) | 49.0 (10.3) | 62.0 | 40.7 (9.9) | 44.2 (11.2) | 37.7 (7.1) | 58.5 (10.6) | 45.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 22 | 0 | 2 | 5 | 1 | 1 | 1 | 1 | 0 | 0 | 38
  Male | 2 | 2 | 2 | 4 | 29 | 4 | 5 | 3 | 5 | 0 | 6 | 5 | 3 | 2 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 48 | 4 | 7 | 8 | 6 | 1 | 6 | 6 | 3 | 2 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 6 | 50 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 51 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2 | 110

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Complete response (CR) is defined as the disappearance of all clinical evidence of disease. Partial response (PR) is a 50% or greater decrease in the sum of the products of perpendicular diameters of all measurable lesions for at least one month. No new lesions may appear, and none may increase. Minor response (MR) is a 25-49% decrease in the sum of the products of the perpendicular diameters of all measurable lesions. Appearance of new lesions following a PR or CR are considered relapses. Patients with progressive disease (PD) and no evidence of stable disease will be taken off study after receiving IL-2.
Time Frame: Every three to four weeks after the treatment, for up to 5 years.
Measure: Number; unit: Participants
Arm/Group | Abl Cells IV + Cyclophosphamide 30 mg/kg | Abl Cells IV + Cyclophosphamide 60 mg/kg | Abl Cells IV+Low Dose IV IL-2 (Initial) | Abl Cells IV+High Dose IV IL-2 (Initial) | Abl Cells IV + MTD IL-2 | Abl Cells IA + MTD (Prior Cells IV on 6) | Abl Cells IA + MTD IL-2 | Abl Cells IA+MTD IL-2 (MART-1 Reactive) | Abl Cells IV + MTD IL-2 no GCSF | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) | Abl Cells IV + SQ IL-2 With GCSF | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 50 | 4 | 6 | 8 | 6 | 1 | 7 | 6 | 3 | 2
Participants
  Complete Response | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 0
  Minor Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  No Response | 3 | 3 | 3 | 6 | 32 | 4 | 5 | 5 | 4 | 0 | 5 | 3 | 2 | 2
  Stable Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 10.5 months
Measure: Number; unit: Participants
Arm/Group | Abl Cells IV + Cyclophosphamide 30 mg/kg | Abl Cells IV + Cyclophosphamide 60 mg/kg | Abl Cells IV+Low Dose IV IL-2 (Initial) | Abl Cells IV+High Dose IV IL-2 (Initial) | Abl Cells IV + MTD IL-2 | Abl Cells IA + MTD (Prior Cells IV on 6) | Abl Cells IA + MTD IL-2 | Abl Cells IA+MTD IL-2 (MART-1 Reactive) | Abl Cells IV + MTD IL-2 no GCSF | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) | Abl Cells IV + SQ IL-2 With GCSF | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 51 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2
Participants | 3 | 3 | 3 | 6 | 50 | 4 | 7 | 8 | 6 | 1 | 7 | 6 | 3 | 2

ADVERSE EVENTS:
Groups:
- Abl Cells IV + SQ IL-2 With GCSF: Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + granulocyte colony stimulating factor (G-CSF) (to shorten time to neutrophil recovery), reactivity not specified
- Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive): Abl Cells intravenous (IV) + subcutaneous (SQ) interleukin-2 (IL-2) with granulocyte colony stimulating factor (GCSF) (melanoma-associated antigen recognized by T cells (MART-1) reactive) Phase 2 Fludarabine 5x25mg/m^2 + Cyclophosphamide 2x60mg/kg + Cells IV + SQ IL-2 (125,000 IU/kg/dose for 5 days for six weeks with 2 days rest per week) + G-CSF + MART-1:26-35(27L) Peptide 1mg/day (5-8 days) in patients with MART-1 reactive cells
Arm/Group | Abl Cells IV + Cyclophosphamide 30 mg/kg | Abl Cells IV + Cyclophosphamide 60 mg/kg | Abl Cells IV+Low Dose IV IL-2 (Initial) | Abl Cells IV+High Dose IV IL-2 (Initial) | Abl Cells IV + MTD IL-2 | Abl Cells IA + MTD (Prior Cells IV on 6) | Abl Cells IA + MTD IL-2 | Abl Cells IA+MTD IL-2 (MART-1 Reactive) | Abl Cells IV + MTD IL-2 no GCSF | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) | Abl Cells IV + SQ IL-2 With GCSF | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 9/51 | 0/4 | 2/7 | 1/8 | 0/6 | 0/1 | 0/7 | 0/6 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 50/51 | 4/4 | 7/7 | 8/8 | 6/6 | 1/1 | 7/7 | 6/6 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Abl Cells IV + Cyclophosphamide 30 mg/kg (N=3) | Abl Cells IV + Cyclophosphamide 60 mg/kg (N=3) | Abl Cells IV+Low Dose IV IL-2 (Initial) (N=3) | Abl Cells IV+High Dose IV IL-2 (Initial) (N=6) | Abl Cells IV + MTD IL-2 (N=51) | Abl Cells IA + MTD (Prior Cells IV on 6) (N=4) | Abl Cells IA + MTD IL-2 (N=7) | Abl Cells IA+MTD IL-2 (MART-1 Reactive) (N=8) | Abl Cells IV + MTD IL-2 no GCSF (N=6) | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) (N=1) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) (N=7) | Abl Cells IV + SQ IL-2 With GCSF (N=6) | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) (N=3) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity) (N=2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection/Febrile neutropenia (infection without neutropenia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abl Cells IV + Cyclophosphamide 30 mg/kg (N=3) | Abl Cells IV + Cyclophosphamide 60 mg/kg (N=3) | Abl Cells IV+Low Dose IV IL-2 (Initial) (N=3) | Abl Cells IV+High Dose IV IL-2 (Initial) (N=6) | Abl Cells IV + MTD IL-2 (N=51) | Abl Cells IA + MTD (Prior Cells IV on 6) (N=4) | Abl Cells IA + MTD IL-2 (N=7) | Abl Cells IA+MTD IL-2 (MART-1 Reactive) (N=8) | Abl Cells IV + MTD IL-2 no GCSF (N=6) | Abl Cells IV+MTD IL-2 no GCSF(gp100 Reactive) (N=1) | Abl Cells IV+MTD IL-2 no GCSF (MART-1reactive) (N=7) | Abl Cells IV + SQ IL-2 With GCSF (N=6) | Abl Cells IV + SQ IL-2 With GCSF (MART-1 Reactive) (N=3) | Abl Cells IV + SQ IL-2 With GCSF (no Reactivity) (N=2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 3 (4) | 4 (5) | 37 (50) | 3 (3) | 5 (8) | 6 (9) | 2 (3) | 1 (1) | 5 (10) | 3 (3) | 1 (1) | 1 (1)
Leukocyte count decreased (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (4) | 6 (7) | 50 (66) | 4 (4) | 5 (8) | 7 (12) | 6 (9) | 1 (1) | 7 (9) | 6 (7) | 3 (3) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 3 (6) | 5 (9) | 50 (80) | 3 (4) | 6 (12) | 8 (19) | 5 (12) | 1 (1) | 7 (13) | 6 (10) | 3 (3) | 2 (4)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (3) | 6 (7) | 50 (70) | 4 (4) | 5 (10) | 7 (11) | 6 (8) | 1 (1) | 7 (8) | 6 (8) | 3 (3) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 16 (19) | 1 (1) | 3 (4) | 6 (6) | 3 (3) | 0 (0) | 3 (7) | 2 (2) | 2 (2) | 1 (1)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 16 (17) | 1 (1) | 2 (4) | 4 (4) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (11) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 11 (12) | 0 (0) | 4 (4) | 4 (4) | 1 (2) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 20 (26) | 1 (1) | 2 (6) | 4 (6) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 23 (27) | 1 (1) | 6 (9) | 5 (5) | 2 (3) | 0 (0) | 4 (5) | 6 (6) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
INR increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (18) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (10) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (15) | 0 (0) | 1 (7) | 3 (5) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter-related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low urine output (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No